CLINICAL TRIAL: NCT02046902
Title: Developing and Testing a Personalized Evidence-based Shared Decision-making Tool for Stent Selection
Acronym: DECIDE-PCI
Status: Completed | Type: Observational
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, John A. Spertus, Daniel Lauer/Missouri Endowed Chair, University of Missouri, Kansas City
Other Study IDs: CE-1304-6448
Record Dates: First submitted 2014-01-22; First posted 2014-01-28 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Heart Diseases
Keywords: coronary artery disease; cardiac stent; PCI procedure; Patient preference
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease; Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Heart disease: Adults with a diagnosis of coronary artery disease and may have had a percutaneous coronary intervention.
- Healthy adults: Adults without a diagnosis of coronary artery disease. Focus groups will be held.

SUMMARY:
The goal of this study is to gather input from patients who have undergone PCI, their family and/or caregivers, and clinicians to develop a patient decision aid. The purpose of the decision aid is to deliver information, including individualized estimates of patients' restenosis risk, in an understandable format that would be informative and assist in decision-making for patients undergoing PCI.

DETAILED DESCRIPTION:
Study Plan: Qualitative research methods (focus groups) will be used to gather the information that would be helpful in decision making as well as review several possible output formats. Several sets of focus groups will be convened, with particular attention to recruitment of a diverse population, including women and underserved minority groups.

Study Procedure: We will gather input to create a clinically useful format for presenting the risk estimates for desired outcomes and support clinical decision-making.

Subjects: We anticipate 2 or 3 patient focus groups of 6-8 individuals and 2 clinician focus groups of 3-5 individuals will be scheduled. Fliers will be posted to enlist potential patients. If necessary, patients will also be contacted by a Cardiovascular Research Coordinator and invited to attend a scheduled focus group. After receiving patient/family/caregiver input, selected clinicians from the Saint Lukes Hospital Staff, including cardiologists, cardiac nurses and other cardiology staff, will be invited to attend a scheduled focus group. The invitation will be sent via email and followed up with a phone call, if necessary. If a clinician focus group is unable to be scheduled, then individual interviews will be conducted.

Setting: Patient and Clinician focus group sessions will be held at Saint Luke's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* English or Spanish speaking
* Presence of coronary disease, or a caregiver/relative of one with coronary disease

Exclusion Criteria:

* non-English or non-Spanish speaking
* dementia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with and without coronary artery disease
Sampling Method: Probability Sample
Enrollment: 586 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Spertus, MD, MPH, Principal Investigator — University of Missouri, Kansas City
Locations (2):
- United States (2):
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Undecided
We would be happy to collaborate with others to run analyses, but do not plan on freely distributing our data. You can see my editorial in CCQO to understand my concerns.

REFERENCES:
- [Derived] Chhatriwalla AK, Decker C, Gialde E, Catley D, Goggin K, Jaschke K, Jones P, deBronkart D, Sun T, Spertus JA. Developing and Testing a Personalized, Evidence-Based, Shared Decision-Making Tool for Stent Selection in Percutaneous Coronary Intervention Using a Pre-Post Study Design. Circ Cardiovasc Qual Outcomes. 2019 Feb;12(2):e005139. doi: 10.1161/CIRCOUTCOMES.118.005139. PMID 30764654
- [Derived] Qintar M, Chhatriwalla AK, Arnold SV, Tang F, Buchanan DM, Shafiq A, Pokharel Y, deBronkart D, Ashraf JM, Spertus JA. Beyond restenosis: Patients' preference for drug eluting or bare metal stents. Catheter Cardiovasc Interv. 2017 Sep 1;90(3):357-363. doi: 10.1002/ccd.26946. Epub 2017 Feb 7. PMID 28168845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2014 and December 2016, patients were recruited from 2 percutaneous coronary intervention (PCI) centers, Saint Luke's Mid America Heart Institute (MAHI) and Truman Medical Center (TMC), following institutional review board (IRB) approval at each site.
Groups:
- Pre-Implementation: Patients who undergo coronary angiography and possible percutaneous coronary intervention (PCI) received an Patient Risk Information Systems Manager (ePRISM) consent form with personalized risk estimates for mortality, bleeding, and target vessel revascularization (TVR) with bare-metal stents (BMS) and drug-eluting stents (DES), but neither the shared decision-making (SDM) tool nor decision coaching.
- Post-implementation With Decision Coaching: Patients received the consent form, the SDM tool for stent selection, and decision coaching
- Post-implementation Without Decision Coaching: Patients received the consent form and the SDM tool, but no decision coaching
Period: Overall Study
Arm/Group | Pre-Implementation | Post-implementation With Decision Coaching | Post-implementation Without Decision Coaching
Started | 336 | 113 | 137
Completed | 336 | 113 | 137
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Implementation | Post-implementation With Decision Coaching | Post-implementation Without Decision Coaching | Total
Number analyzed (Participants) | 336 | 113 | 137 | 586
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number analyzed for this baseline measure reflects data captured and does account for missing or unknown data.
  years
    number analyzed (Participants) | 333 | 113 | 137 | 583
    (all) | 66.1 (11.8) | 67.6 (12.9) | 68.6 (11.6) | 67.43 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed for this baseline measure reflects data captured and does account for missing or unknown data.
  Participants
    number analyzed (Participants) | 259 | 110 | 137 | 506
    Female | 93 | 39 | 49 | 181
    Male | 166 | 71 | 88 | 325
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed for this baseline measure reflects data captured and does account for missing or unknown data.
  Participants
    number analyzed (Participants) | 327 | 112 | 135 | 574
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 77 | 21 | 18 | 116
    White | 250 | 91 | 116 | 457
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Number analyzed for this baseline measure reflects data captured and does account for missing or unknown data.
  Participants
    Hispanic Ethnicity: number analyzed (Participants) | 291 | 112 | 132 | 535
    Hispanic Ethnicity | 5 | 2 | 3 | 10
Site [Count of Participants; unit: Participants]
  Mid America Heart Insitute | 191 | 86 | 132 | 409
  Truman Medical Center/Univ. of Missouri KC | 145 | 27 | 5 | 177
Diabetes [Count of Participants; unit: Participants] — Population: Number analyzed for this baseline measure reflects data captured and does account for missing or unknown data.
  Participants
    number analyzed (Participants) | 335 | 113 | 131 | 579
    (all) | 152 | 49 | 69 | 270
Hypertension [Count of Participants; unit: Participants] | 266 | 92 | 106 | 464
Peripheral arterial disease [Count of Participants; unit: Participants] — Population: Number analyzed for this baseline measure reflects data captured and does account for missing or unknown data.
  Participants
    number analyzed (Participants) | 331 | 113 | 121 | 565
    (all) | 29 | 22 | 20 | 71
Prior Coronary Artery Bypass Graft [Count of Participants; unit: Participants] — Population: Number analyzed for this baseline measure reflects data captured and does account for missing or unknown data.
  Participants
    number analyzed (Participants) | 334 | 113 | 127 | 574
    (all) | 53 | 20 | 28 | 101
Prior Percutaneous Coronary Intervention [Count of Participants; unit: Participants] — Population: Number analyzed for this baseline measure reflects data captured and does account for missing or unknown data.
  Participants
    number analyzed (Participants) | 333 | 113 | 133 | 579
    (all) | 137 | 50 | 66 | 253
Admission Status [Count of Participants; unit: Participants] — Population: Number analyzed for this baseline measure reflects data captured and does account for missing or unknown data.
  Participants
    number analyzed (Participants) | 326 | 111 | 129 | 566
    Inpatient | 116 | 44 | 57 | 217
    Outpatient | 189 | 67 | 71 | 327
    Emergent | 21 | 0 | 1 | 22

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Pre-implementation, Post-implementation With Decision Coaching, and Post-implementation Without Decision Coaching
Description: The primary outcome was whether or not patients participated in SDM regarding stent choice. Patients were categorized as having participated in SDM if they answered anything other than "doctor alone" in response to the question "Who chose the type of stent?"
Time Frame: 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation | Post-implementation With Decision Coaching | Post-implementation Without Decision Coaching
Number analyzed (Participants) | 336 | 113 | 137
Participants
  Doctor Alone | 235 | 45 | 106
  Mostly Doctor | 51 | 19 | 20
  Doctor and you equally | 40 | 32 | 4
  Mostly you | 2 | 11 | 6
  You alone | 8 | 6 | 1

2. Secondary Outcome: Concordance Between Stent Preference and Stent Received Was a Secondary Outcome.
Description: Secondary outcomes included patients' recall of individual aspects of the stent discussion, stent knowledge score, patient preference for stent type, perceived autonomy support from their providers ,and concordance of patient stent preference and type of stent received. Patients were categorized as having voiced a stent preference if they answered anything other than "I don't care" or "I don't know" in response to the question "After reviewing the risks and benefits of both types of stents, which type of stent did you want?"
Time Frame: 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Implementation | Post-implementation With Decision Coaching | Post-implementation Without Decision Coaching
Number analyzed (Participants) | 336 | 113 | 137
Participants
  Drug eluting stent | 83 | 49 | 23
  Bare metal stent | 36 | 29 | 2
  I don't care | 119 | 29 | 69
  I don't know | 98 | 6 | 43

ADVERSE EVENTS:
Description: There was not a Data Safety Monitoring Board as this was deemed low risk and no Serious, and Other [Not Including Serious] Adverse Events were monitored/recorded.
Arm/Group | Pre-Implementation | Post-implementation With Decision Coaching | Post-implementation Without Decision Coaching
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The lack of randomization, availability of ePrism at hospitals, estimation of TVR risk in the SDM tool without the availability of angiographic data, and physicians were not surveyed for additional variables that impacted their stent selection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No